CLINICAL TRIAL: NCT04259203
Title: Efficacy of Ericksonian Hypnosis in the Management of Chronic Pain Related to Parkinson's Disease
Acronym: DOLHYP-PARK-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: France Parkinson Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-51; 2019-A00539-48 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2022-05

CONDITIONS: Parkinson Disease; Chronic Pain
Keywords: No-motor symptoms; Pain perception; Quality of life; Hypnosis; Auto-hypnosis
MeSH Terms: conditions — Parkinson Disease; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erickson hypnosis (Experimental): 5 sessions of Erickson hypnosis (1 session per week), associated with autohypnosis at home in-between sessions.
  Interventions: Behavioral: Erickson hypnosis
- Usual care (No Intervention): Usual management of pain symptoms

INTERVENTIONS:
Behavioral: Erickson hypnosis — Erickson hypnosis sessions performed by an experienced hypnotherapist, according to a pre-established protocol : 5 sessions (1 per week). Between each session : exercise of auto-hypnosis by the patient himself, at home
  Arms: Erickson hypnosis

SUMMARY:
This study evaluates the efficacity of Erickson hypnosis in the treatment of chronic pain in patients with Parkinson's disease. Half of participants will follow a 2-month Erickson hypnosis protocole, while the other half will benefit from the usual care.

DETAILED DESCRIPTION:
A large proportion of patients with Parkinson's disease suffer of chronic pain directly related to the disease. The management of painful symptoms is difficult and currently, there is no commonly admitted guidelines.

Several studies have shown the efficacy of Erickson hypnosis to reduce the perception of chronic pain in different conditions. This efficacy has never been tested in Parkinson's disease.

The objective of this study is to assess the efficacy of Erickson hypnosis protocol, compared to usual care, for the management of Parkinson's disease-related chronic pain.

The study team assume that Erickson hypnosis will be more efficient than usual care to reduce perceived chronic pain. They also assume that regular practice of autohypnosis will contribute to long-term efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Men or women
* 18 to 80 years old
* idiopathic Parkinson's disease
* without neurological co-morbidity
* Suffering from chronic pain (for at least 3 months), related to Parkinson's disease
* Having a pain intensity of at least 30 mm on the VAS (average intensity over the previous week) for Parkinson's disease-related pain
* antiparkinsonian, analgesic and psychotropic treatments stable for 1-month
* having a health insurance
* signed informed consent form

Exclusion Criteria:

* Patient with a neurological condition other than Parkinson's disease or with an atypical Parkinson's syndrome
* Early untreated patient
* Patient with acute intercurrent pain
* Patient whose pain is mainly attributable to another pathology (rheumatoid arthritis, spondyloarthritis ankylosing, diabetic neuropathy, cancer, etc.)
* Patient with cognitive impairment objectified by a score at the Montreal Cognitive Assessment (MoCA) <24
* Patient with hallucinations and/or psychosis (MDS-UPDRS 1.2> 1)
* Patient with a apathy (MDS-UPDRS 1.5> 1)
* Patient with disabling dyskinesia (MDS-UPDRS) 4.1 AND 4.2> 1)
* Patient under the protection of adults
* Pregnant or lactating woman

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-08-08 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2024-08-16 (Actual)

PRIMARY OUTCOMES:
Change of the intensity of pain perception | At baseline and 2 months after
  Measure of the intensity of pain perception by VAS at the baseline visit and at the post-treatment visit (2 months later). The difference between both values will allow to calculate a variation index.

SECONDARY OUTCOMES:
Change of the score at the Brief Pain Inventory | At baseline and 2 months after
  Completion of the Brief Pain Inventory at the baseline visit and at the post-treatment visit (2 months later). The difference between both scores will allow to calculate a variation index.
Change of the score at the McGill Pain Questionnaire | At baseline and 2 months after
  Completion of the McGill Pain Questionnaire at the baseline visit and at the post-treatment visit (2 months later). The difference between both scores will allow to calculate a variation index.
Change of the score at the Beck Depression Inventory | At baseline and 2 months after
  Completion of the Beck Depression Inventory at the baseline visit and at the post-treatment visit (2 months later). The difference between both scores will allow to calculate a variation index.
Change of the score at the Fatigue Severity Scale | At baseline and 2 months after
  Completion of the Fatigue Severity Scale at the baseline visit and at the post-treatment visit (2 months later). The difference between both scores will allow to calculate a variation index.
Change of the score at the Parkinson's Disease Questionnaire-8 (PDQ-8) | At baseline and 2 months after
  Completion of the PDQ-8 at the baseline visit and at the post-treatment visit (2 months later). The difference between both scores will allow to calculate a variation index.
Change of the score at the Scale for Outcomes at Parkinson's Disease (SCOPA-PS) | At baseline and 2 months after
  Completion of the SCOPA-PS at the baseline visit and at the post-treatment visit (2 months later). The difference between both scores will allow to calculate a variation index.
Change of the score at the Euroqol 5 dimensions 5 levels (EQ-5D-5L) | At baseline and 2 months after
  Completion of the EQ-5D-5L at the baseline visit and at the post-treatment visit (2 months later). The difference between both scores will allow to calculate a variation index.
Change in the dose of analgesic treatments | At baseline and 2 months after
  Analgesic treatments will be recorded during the week preceding each visit and a mean dosage will be calculated during each period. The difference between both mean values will allow to calculate a variation index.
Change in the dose of psychotropic medications | At baseline and 2 months after
  Psychotropic medications will be recorded during the week preceding each visit and a mean dosage will be calculated during each period. The difference between both mean values will allow to calculate a variation index.
Change of the score at MDS-UPDRS | At baseline and 2 months after
  Completion of the MDS-UPDRS at the baseline visit and at the post-treatment visit (2 months later). The difference between both scores will allow to calculate a variation index.

CONTACTS AND LOCATIONS:
Overall Officials: Luc Defebvre, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (4):
- France (4):
  - Chu Cote de Nacre, Caen
  - Hôpital Roger Salengro, CHRU de Lille, Lille
  - Hopital Charles Nicolle Chu Rouen, Rouen
  - Hopital Purpan Chu Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No